CLINICAL TRIAL: NCT03086863
Title: Effectiveness and Safety of Electroacupuncture for Poststroke Patients With Shoulder Pain: Study Protocol for a Multicenter, Randomized, Patient and Assessor Blinded, Sham Controlled, Parallel, Clinical Trial
Brief Title: Electroacupuncture for Poststroke Patients With Shoulder Pain
Acronym: EAPSSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyunghee University (Other)
Collaborators: Wonkwang University Gwangju Medical Center (Unknown); National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Lee Eui-ju, Professor, Ph.D. KMD., Kyunghee University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017005
Record Dates: First submitted 2017-02-26; First posted 2017-03-22 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Stroke; Shoulder Pain; Stroke, Complication; Cerebral Infarction; Cerebral Hemorrhage
Keywords: electroacupuncture; randomized controlled trial
MeSH Terms: conditions — Stroke; Shoulder Pain; Cerebral Infarction; Cerebral Hemorrhage | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- verum electroacupuncture (Experimental): * Electroacupuncture on LI4, LI15, TE14, SI9, SI11, and GB21, unilaterally
  * Needle insertion by 10-15 mm and de qi sensation
  * Park sham guide tubes
  * Low frequency electronic stimulation (30 Hz)
  * Retention for 20 minutes.
  Interventions: Device: electroacupuncture
- sham electroacupuncture (Sham Comparator): * Park sham device on on LI4, LI15, TE14, SI9, SI11, and GB21, unilaterally
  * Needle installation without penetration
  * Park sham guide tubes
  * Low frequency electronic stimulation (30 Hz) for a fake noise without conduction
  * Retention for 20 minutes.
  Interventions: Device: sham electroacupuncture

INTERVENTIONS:
Device: electroacupuncture — All the patients in verum electroacupuncture group will receive acupuncture on the six adjacent acupoints (LI4, LI15, TE14, SI9, SI11, and GB21) in unilateral side. Acupuncture needles (stainless steel, 0.25 mm × 40 mm, Dong Bang Acupuncture Inc., Republic of Korea) will be inserted 10-15 mm in depth and de qi sensation will be elicited. Park sham guide tubes will be used in verum group, too. Low frequency stimulate (STN-111, Stratek, Republic of Korea) will be connected to the tips of needles to provide electrical stimulation at middle frequency (30 Hz). Needles with electrical stimulation will be retained for 20 minutes. Patients should take this procedure 3 times a week for 3 weeks (9 sessions in total).
  Other Names: verum EA
  Arms: verum electroacupuncture
Device: sham electroacupuncture — We selected a non-penetrating sham needling, i.e., Park sham device, which has been developed and validated in preceding studies as comparison. On the exactly same 6 acupoints as verum electroacupuncture group, needles will be installed with Park sham guide tubes and the same electrical stimulators will be connected the tips of needles. Since the needles do not penetrate the skin, the stimulation is not electrically conducted. To be sure of patient blinding, the low frequency stimulate will be turned on with the same frequency (30 Hz), which makes a fake noise, resulting in letting patients believe that they are taking real electroacupuncture therapy for 20 minutes. Sham group will also 9 session for 3 weeks (3 sessions a week).
  Other Names: sham EA
  Arms: sham electroacupuncture

SUMMARY:
This is a multicenter, randomized, sham-controlled, patient- and assessor-blinded, and parallel trial to explore the effectiveness and safety of electroacupuncture (EA) therapy, compared with sham EA, for poststroke shoulder pain.

DETAILED DESCRIPTION:
This study is aimed at showing the effectiveness and safety of electroacupuncture therapy for the stroke survivors with shoulder pain. 60 stroke survivors with shoulder pain will be enrolled in two traditional Korean medicine hospitals and randomly divided into either of verum or sham electroacupuncture group with 1:1 of allocation ratio. The participants will receive 9 sessions of electroacupuncture procedures for 3 weeks. Patients and outcome assessors will be blinded from the beginning to the study completion. Visual analogue scale will be primarily evaluated, and pain rating scale, Fugl-Meyer assessment upper extremity, modified Ashworth scale, manual muscle test, passive range of motion, Korean version of modified Barthel index, and Korean version of Beck depression inventory will be measured, too. Blinding index will be assessed. For safety, adverse events will be collected.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with cerebral hemorrhage or infarction examined by computed tomography (CT) magnetic resonance imaging (MRI) at least 2 weeks or more ago;
* complaining hemiplegic shoulder pain of VAS ≥4;
* agreeing that any treatments, including analgesics, for hemiplegic shoulder pain will not be changed from the previous 2 weeks prior to the enrollment until the last evaluation, if applicable;
* fully explained about the clinical research and sign the informed consents.

Exclusion Criteria:

* disorders, traumatic injury, or surgery of shoulders even before their stroke;
* pacemakers, embedded neural stimulator, cardiac arrhythmia, epilepsy, peripheral neural injury on their medical history;
* psychiatric disorders;
* cancer within the past 5 years, regardless of its prognosis and location;
* cognitive impairment that interferes with clinical assessment;
* hypersensitivity or fears to acupuncture;
* bleeding disorders (e.g. hemophilia or von Willebrand disease, etc.),
* pregnancy,
* difficulty in communicating with researchers, or
* any other conditions who are considered inappropriate for participating in the trial by experienced practitioners.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Mean difference of visual analogue scale (VAS) between baseline and endpoint | 3 weeks
  VAS is a patient-rated outcome with a 10-cm line representing 'not painful at all' for zero and 'most painful' for ten. Patient marks x on the line by oneself, based on how intense he/she thinks the pain is and assessor measures the length from zero point to x mark, which is the pain score.

SECONDARY OUTCOMES:
before-after change of visual analogue scale (VAS) (intragroup effect) | 1~3 weeks
  VAS is a patient-rated outcome with a 10-cm line representing 'not painful at all' for zero and 'most painful' for ten. Patient marks x on the line by oneself, based on how intense he/she thinks the pain is and assessor measures the length from zero point to x mark, which is the pain score.
Mean difference of pain rating scale (PRS) between baseline and endpoint | 3 weeks
  PRS is a patient-rated outcome to assess pain with 4 items for intensity (0-10 points), frequency (0-5 points), duration (0-5 points) and aggravating factors (0-5 points). The pain score is the product of the intensity point and the sum of frequency, duration, aggravating factors points (0-150 points in total).
Mean difference of Fugl-Meyer assessment - upper extremity (FMA-UE) between baseline and endpoint | 3 weeks
  FMA-UE assesses physical performance of upper extremity following stroke. The original FMA scale includes 4 domains of motor function, sensation qualities, passive range of motion, and joint pain with 3-point items ('cannot perform' for 0, 'perform partially' for 1, and 'perform fully' for 2). We are going to measure only 8 items for upper extremity (shoulder retraction, elevation, abduction, abduction to 90°, adduction/internal rotation, external rotation, flexion 0-90°, and flexion 90-180°)
Mean difference of passive ranges of motion (PROM) between baseline and endpoint | 3 weeks
  PROM for shoulder flexion, abduction, and extension will be measured with goniometer. The maximum degrees under passive movement of shoulder unless patients suffer from pain will be tested.
Mean difference of manual muscle test (MMT) between baseline and endpoint | 3 weeks
  MMT assesses muscle strength in poststroke shoulder injury. Assessors will rate on a grade of 0 (no contraction at all) to 5 (complete range of motion against gravity with maximum resistance) for hemiplegic shoulder.
Mean difference of modified Ashworth scale (MAS) between baseline and endpoint | 3 weeks
  MAS is a clinical rating scale to measure tonal abnormality after stroke. Assessors should grade from 0, meaning no increase in muscle tone, to 5, meaning that rigid shoulder on flexion or extension.
Mean difference of Korean version of modified Barthel index (K-MBI) between baseline and endpoint | 3 weeks
  K-MBI is an ordinal scale used to measure performance in activities of daily living. Ten items (personal hygiene, bathing, feeding, toilet use, stair climbing, dressing, bowel control, bladder control, walking, and chair/bed transfers) will be graded between 1 (completely dependent on others to perform) and 5 (completely independent on others to perform), respectively, and it scores up to 100 points in total.
Mean difference of Korean version of Beck depression inventory (K-BDI) between baseline and endpoint | 3 weeks
  K-BDI is a patient-rated outcome with 21 items, 0 to 3 points of each item. The higher the total score is, the severe the depressive level is.
mean difference of the occurrence numbers of adverse events | 3 times per week, 3 weeks, through study completion,
  At every visit, assessors will ask a post-interventional question about adverse events. The number of adverse events will be recorded for each group.

OTHER OUTCOMES:
new Blinding index (BI) | 3 weeks (only at the end of the study)
  Patients and outcome assesses will be asked which group they think they belong to and select one of the answers (verum electroacupuncture group, sham electroacupuncture group, or unknown). With the answers, the new BI will be calculated with mean and variances following the preceding study. The index score varies from 1 of complete lack of blinding, 0 of consistency with perfect blinding, or -1 of opposite guessing of their groups.

CONTACTS AND LOCATIONS:
Overall Officials: Euiji Lee, Ph.D., Principal Investigator — Kyunghee University
Locations (1):
- Kyung Hee University Korean Medicine Hospital, Seoul, South Korea

REFERENCES:
- [Background] Lee SH, Lim SM. Acupuncture for Poststroke Shoulder Pain: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2016;2016:3549878. doi: 10.1155/2016/3549878. Epub 2016 Jul 31. PMID 27547224
- [Background] Bang H, Ni L, Davis CE. Assessment of blinding in clinical trials. Control Clin Trials. 2004 Apr;25(2):143-56. doi: 10.1016/j.cct.2003.10.016. PMID 15020033
- [Background] Park J, White A, Stevinson C, Ernst E, James M. Validating a new non-penetrating sham acupuncture device: two randomised controlled trials. Acupunct Med. 2002 Dec;20(4):168-74. doi: 10.1136/aim.20.4.168. PMID 12512790
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Kim C, Kim C, Chun SI. Clinical value of a new self assessment method of pain. Journal of Korean Acamedy of Rehabilitation Medicine 22(2):305-311, 1998. (Korean)
- [Background] Kim HS, Her JG, Ko JY, Park DS, Woo JH, You YY, Choi YE. Reliability, concurrent validity, and responsiveness of the Fugl-Meyer assessment (FMA) for hemiplegic patients. Journal of Physical Therapy Science 24(9):893-899, 2012.
- [Background] Mendell JR, Florence J. Manual muscle testing. Muscle Nerve. 1990;13 Suppl:S16-20. doi: 10.1002/mus.880131307. No abstract available. PMID 2233877
- [Background] Gregson JM, Leathley M, Moore AP, Sharma AK, Smith TL, Watkins CL. Reliability of the Tone Assessment Scale and the modified Ashworth scale as clinical tools for assessing poststroke spasticity. Arch Phys Med Rehabil. 1999 Sep;80(9):1013-6. doi: 10.1016/s0003-9993(99)90053-9. PMID 10489001
- [Background] Jung HY, Park BK, Shin HS, Kang YK, Pyun SB, Paik NJ, Kim SH, Kim TH, Han TR. Development of the Korean version of modified barthel index (K-MBI): multi-center study for subjects with Stroke. Journal of Korean Acamedy of Rehabilitation Medicine 31(3):283-297, 2007. (Korean)
- [Background] Rhee MK, Lee YH, Park SH, Sohn CH, Chung YC, Hong SK, Lee BK, Chang P, Yoon AR. A stadardization study of beck depression inventory Ⅰ - Korean version (K-BDI): reliability and factor analysis. The Korean Journal of Psychopathology 4(1):77-95, 1995. (Korean)
- [Background] Rhee MK, Lee YH, Jung HY, Chio JH, Kim SH, Kim YK, Lee SK. A stadardization study of beck depression inventory Ⅱ - Korean version (K-BDI): validity. The Korean Journal of Psychopathology 4(1):96-104, 1995 . (Korean)
- [Background] Wang KF, Zhang LJ, Lu F, Lu YH, Yang CH. Can Ashi points stimulation have specific effects on shoulder pain? A systematic review of randomized controlled trials. Chin J Integr Med. 2016 Jun;22(6):467-72. doi: 10.1007/s11655-015-2107-4. Epub 2015 Jun 30. PMID 26129899
- [Derived] Shin S, Yang SP, Yu A, Yoo J, Lim SM, Lee E. Effectiveness and safety of electroacupuncture for poststroke patients with shoulder pain: study protocol for a double-center, randomized, patient- and assessor-blinded, sham-controlled, parallel, clinical trial. BMC Complement Altern Med. 2019 Mar 12;19(1):58. doi: 10.1186/s12906-019-2468-x. PMID 30866914